CLINICAL TRIAL: NCT01448642
Title: A Randomized, Multicenter Clinical Trial to Assess the Effect of Atorvastatin in Patients With Acute Coronary Syndrome and Intended Percutaneous Coronary Intervention
Brief Title: Statins Evaluation in Coronary Procedures and Revascularization Trial
Acronym: SECURE-PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 185/2011
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin loading dose of 80mg before PCI, reloading dose of 80mg 24 hours after PCI, and atorvastatin 40mg for 30 days
  Arms: Atorvastatin
Drug: Placebo — Matching placebo before PCI and 24 hours after PCI. Atorvastatin 40mg for 30 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a loading dose of atorvastatin before percutaneous intervention procedures in acute coronary syndromes is effective to reduce major cardiovascular events(MACE).

DETAILED DESCRIPTION:
Background: Strategies to reduce complications in acute coronary syndrome treatment have been largely studied. Due to its pleiotropic effects statins are considered an important tool on atherosclerotic plaque stability. Although, the usage of statins before percutaneous coronary intervention in acute coronary syndrome patients, has not yet been demonstrated. Objectives: Evaluate if a loading dose of atorvastatin (80mg) before percutaneous coronary intervention in acute coronary syndrome patients, followed by a reload dose 24 hours, is able to reduce major cardiovascular events (MACE); including combined outcomes such as all-cause mortality, nonfatal acute myocardial infarction, stroke or revascularization with either percutaneous coronary intervention or coronary-artery bypass grafting after 30 days. Methods: Multicentric randomised controlled clinical trial, with allocation concealment and intention to treat analysis. Competitive recruitment will involve 4,192 patients. Acute coronary syndrome patients intending to undergo percutaneous coronary intervention with or without stent placement will be randomized 1:1 to receive either atorvastatin 80mg or placebo before the coronary procedure and also a reload dosage after 24 hours from angioplasty. All patients will collect blood sample to determine CKMB levels pre and post procedure (6 to 12h and 18 to 24 hours). After 30 days, an in person interview will be performed and blood sample will be collected in order to dosage AST, ALT, CPK, and cholesterol levels. Telephonic interview will be done at 6 and 12 months to access occurrence of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome patients intending to undergo percutaneous coronary intervention.

Exclusion Criteria:

* Younger than 18 years
* Presence of any contraindication to statin (Pregnant women, breast-feeding women or statin hypersensibility)
* Advanced hepatic disease
* Use of statins at the maximum dosage in the last 24 hours before the loading dose of the study drug
* Use of fibrate in the last 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4191 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Major Cardiovascular Events (MACE) | 30 days
  All-cause mortality, nonfatal acute myocardial infarction, stroke or revascularization with either percutaneous coronary intervention or coronary artery bypass grafting

SECONDARY OUTCOMES:
Major Cardiovascular Events (MACE) | 6 months and 12 months
All-cause mortality | 30 days, 6 months and 12 months
Non-fatal Myocardial Infarction | 30 days, 6 months and 12 months
Non-fatal Stroke | 30 days, 6 months and 12 months
Revascularization | 30 days, 6 months and 12 months
Cardiovascular death | 30 days, 6 months and 12 months
Stent Thrombosis | 30 days, 6 months and 12 months
Target vessel revascularization | 30 days, 6 months and 12 months
Rhabdomyolysis | 7 days or at hospital discharge
Bleeding episode | 7 days or hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Otavio Berwanger, Study Chair — Hospital do Coracao; Renato D Lopes, MD, PhD, Study Chair — Brazilian Clinical Research Institute
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Berwanger O, Santucci EV, de Barros E Silva PGM, Jesuino IA, Damiani LP, Barbosa LM, Santos RHN, Laranjeira LN, Egydio FM, Borges de Oliveira JA, Dall Orto FTC, Beraldo de Andrade P, Bienert IRC, Bosso CE, Mangione JA, Polanczyk CA, Sousa AGMR, Kalil RAK, Santos LM, Sposito AC, Rech RL, Sousa ACS, Baldissera F, Nascimento BR, Giraldez RRCV, Cavalcanti AB, Pereira SB, Mattos LA, Armaganijan LV, Guimaraes HP, Sousa JEMR, Alexander JH, Granger CB, Lopes RD; SECURE-PCI Investigators. Effect of Loading Dose of Atorvastatin Prior to Planned Percutaneous Coronary Intervention on Major Adverse Cardiovascular Events in Acute Coronary Syndrome: The SECURE-PCI Randomized Clinical Trial. JAMA. 2018 Apr 3;319(13):1331-1340. doi: 10.1001/jama.2018.2444. PMID 29525821
- [Derived] Lopes RD, de Barros E Silva PGM, de Andrade Jesuino I, Santucci EV, Barbosa LM, Damiani LP, Nakagawa Santos RH, Laranjeira LN, Dall Orto FTC, Beraldo de Andrade P, de Castro Bienert IR, Alexander JH, Granger CB, Berwanger O. Timing of Loading Dose of Atorvastatin in Patients Undergoing Percutaneous Coronary Intervention for Acute Coronary Syndromes: Insights From the SECURE-PCI Randomized Clinical Trial. JAMA Cardiol. 2018 Nov 1;3(11):1113-1118. doi: 10.1001/jamacardio.2018.3408. PMID 30264159
- [Derived] Berwanger O, de Barros E Silva PGM, Dall Orto FTC, de Andrade PB, de Castro Bienert IR, Bosso CE, Mangione J, Polanczyk CA, Sousa A, Kalil R, de Moura Santos L, Sposito AC, Rech RL, Sousa ACS, Baldissera F, Nascimento BR, de Andrade Jesuino I, Santucci EV, Damiani LP, Laranjeira LN, Borges de Oliveira JA, Giraldez RR, Cavalcanti AB, Pereira SB, Mattos LA, Armaganijan LV, Guimaraes HP, Sousa JE, Alexander JH, Granger CB, Lopes RD. Rationale and design of the Statins Evaluation in Coronary procedUres and REvascularization: The SECURE-PCI Trial. Am Heart J. 2018 Apr;198:129-134. doi: 10.1016/j.ahj.2017.12.018. Epub 2018 Jan 8. PMID 29653634